CLINICAL TRIAL: NCT00908765
Title: Effects of Aerobe Interval Training and Moderate Continuous Training in COPD Patients
Brief Title: Effects of Aerobe Interval Training and Moderate Continuous Training in Chronic Obstructive Pulmonary Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 42008754
Record Dates: First submitted 2009-04-20; First posted 2009-05-27 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2013-01

CONDITIONS: COPD; Chronic Obstructive Pulmonary Disease
Keywords: Exercise Training COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aerobe Interval Training (Active Comparator): High aerobic intensity treadmill walking. 4 by 4 minutes interval training on a graded treadmill at a heart rate corresponding to 85-95% of maximal heart rate. 3 times per week for 10 weeks.
  Interventions: Behavioral: Exercise
- Moderate Continous Training (Active Comparator): Moderate continuous intensity treadmill walking on a graded treadmill at a heart rate corresponding to 60-70 of maximal heart rate, 3 times per week for 10 weeks
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — 1. High aerobic intensity treadmill walking. 4 by 4 minutes interval training on a graded treadmill at a heart rate corresponding to 85-95% of maximal heart rate. 3 times per week for 10 weeks.
  2. Moderate continuous intensity treadmill walking on a graded treadmill at a heart rate corresponding to 60-70 of maximal heart rate, 3 times per week for 10 weeks
  Other Names: non

SUMMARY:
Reduced exercise tolerance is one of the hallmarks of COPD. The principal causes for exercise intolerance are ventilatory limitation leading to deconditioning and inactivity. So far it is poorly understood which form of exercise is the most effective in training this condition. The investigators want to study the physiological response to two different training programs (High intensity aerobe interval training and moderate continuous aerobe training)with special focus on cardiac and skeletal muscle adaptions

DETAILED DESCRIPTION:
Reduced exercise tolerance is one of the hallmarks of COPD and The principal causes for exercise intolerance are ventilatory limitation leading to deconditioning and inactivity. However the weak correlation between exercise capacity and FEV1 implies that other factors than reduced pulmonary function contributes to this impairment . Several studies have found changes in skeletal muscle, with fibre shift, increased oxidative stress, increased inflammatory cytokines and impaired mitochondrial function, suggesting a lower limb dysfunction

Numerous exercise studies in COPD patients have shown physiological and physiological benefits of training and endurance training is now regarded as an important part in pulmonary rehabilitation. It is still uncertain what type of endurance training that is most favourable for COPD patients.

In patients with heart failure and metabolic syndrome aerobe interval exercise have be shown to be superior in improving aerobic capacity and cardiac function

We therefore want conduct a study comparing training effects in patients with moderate to severe COPD, that participated in an identical training program that in HF and metabolic syndrome patients gave significant improvement in aerobic capacity, cardiac function and skeletal muscle function.

Patients will therefore be assigned to either 4x4 minutes high intensity interval treadmill exercise or continuous moderate intensity treadmill exercise 3 times pr week for 12 weeks. Aerobic capacity and work economy, pulmonary,cardiac and skeletal muscle function before and after the exercise training will be measured.

ELIGIBILITY:
Inclusion Criteria:

* COPD with FEV1 25-60 % of exp , FEV1%FVC<70 %. Age 45-80 years

Exclusion Criteria:

* Heart failure
* symptomatic coronary artery disease
* cancer
* alcohol and drug abuse
* severe mental illness
* Lower respiratory infection last 4 weeks
* participation in exercise- or lung rehabilitation program last 3 months.
* oral steroid use

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-08; Primary Completion 2008-12 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
VO2-peak | At inclusion and after 12 weeks of exercise training

SECONDARY OUTCOMES:
Cardiac function | At inclusion and after 12 weeks of exercise training
Skeletal muscle function | At inclusion and after 12 weeks of exercise training

CONTACTS AND LOCATIONS:
Overall Officials: Sigurd Steinshamn, MD PhD, Principal Investigator — NTNU , Trondheim; Eivind Brønstad, MD, Principal Investigator — NTNU, Trondheim
Locations (1):
- Department of Circulation and Medical Imaging , NTNU, Trondheim, Trondheim, Norway

REFERENCES:
- [Result] Bronstad E, Tjonna AE, Rognmo O, Dalen H, Heggli AM, Wisloff U, Ingul CB, Steinshamn S. Aerobic exercise training improves right- and left ventricular systolic function in patients with COPD. COPD. 2013 Jun;10(3):300-6. doi: 10.3109/15412555.2012.745843. Epub 2012 Dec 28. PMID 23272664